CLINICAL TRIAL: NCT01240265
Title: Maternal Oral Vitamin D Supplementation Via Daily or Monthly Regimens and the Effect on Levels of Vitamin D in Human Milk and Infant Serum
Brief Title: Vitamin D Supplementation in Breastfeeding Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thomas Thacher, Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-004130
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Vitamin D Deficiency; Rickets; Infant Nutrition Disorders
Keywords: Vitamin D deficiency; Rickets; Infant; Nutrition
MeSH Terms: conditions — Vitamin D Deficiency; Rickets; Infant Nutrition Disorders | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D 150,000 units once (Experimental): Single dose of vitamin D3 150,000 IU given orally once
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D 5000 units daily (Experimental): Vitamin D3 5000 IU daily given orally for 28 days
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 150,000 IU orally given once
  Other Names: Cholecalciferol
  Arms: Vitamin D 150,000 units once
Dietary Supplement: Vitamin D3 — 5000 IU given orally daily for 28 days
  Other Names: Cholecalciferol
  Arms: Vitamin D 5000 units daily

SUMMARY:
Adequate vitamin D is essential for proper infant growth and development. However, human milk is low in vitamin D, and most infants do not receive recommended supplementation. Our aim is to assess the feasibility of providing adequate vitamin D to breastfed infants through maternal vitamin D supplementation. Forty non-pregnant, lactating women at least 18 years of age with exclusively breastfed infants between the ages of 1 and 6 months will be randomized to receive oral vitamin D as either 5,000 IU daily for 28 days or 150,000 IU as a single dose. Maternal serum calcium, phosphorus, vitamin D and 25(OH)D; maternal urinary calcium; maternal milk vitamin D and 25(OH)D will be measured on days 0, 1, 3, 7, 14, and 28 of the study; and infant serum vitamin D and 25(OH)D will be measured on days 0 and 28.

ELIGIBILITY:
Inclusion criteria

* Currently lactating mothers at least 18 years of age
* Willing to continue exclusively breastfeeding their infant throughout the study interval
* The infant is 1-6 months of age at the beginning of the study
* Willing and able to participate in all aspects of the study
* Mother and infant are in good health, as determined by the study investigator
* Have been provided with, understand, and have signed the informed consent for themselves and their child.

Exclusion criteria

* Have recently travelled (within the preceding 30 days) or plan to travel south of 35 degrees north latitude during the study interval
* Have recently or plan to engage in indoor tanning
* Are currently taking medications that affect vitamin D metabolism, like steroids, anticonvulsants, or barbiturates
* Are nursing multiple infants (e.g. twins)
* Are taking greater than the daily recommended intake of 1000 mg elemental calcium as calcium supplements
* Are taking greater than the standard daily dose of 400 IU of vitamin D found in prenatal vitamins
* Infant weight below 1.67 kg
* Mothers with baseline 25(OH)D levels >70 ng/ml, and/or infants with baseline 25(OH)D levels >70 ng/ml
* History of kidney stones

Ages: 1 Month to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The number of days of detectable milk vitamin D concentrations | 28 days
  To compare the number of days of detectable milk vitamin D concentrations and incremental area under the curve between two dosing regimens of oral cholecalciferol in lactating mothers.

SECONDARY OUTCOMES:
Infant serum 25(OH)D concentration | 28 days
  To compare the change in serum 25(OH)D concentrations in infants receiving milk from mothers supplemented with either 5,000 IU daily or 150,000 IU monthly cholecalciferol

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Thacher, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Ketha H, Thacher TD, Oberhelman SS, Fischer PR, Singh RJ, Kumar R. Comparison of the effect of daily versus bolus dose maternal vitamin D3 supplementation on the 24,25-dihydroxyvitamin D3 to 25-hydroxyvitamin D3 ratio. Bone. 2018 May;110:321-325. doi: 10.1016/j.bone.2018.02.024. Epub 2018 Feb 24. PMID 29486367
- [Derived] Oberhelman SS, Meekins ME, Fischer PR, Lee BR, Singh RJ, Cha SS, Gardner BM, Pettifor JM, Croghan IT, Thacher TD. Maternal vitamin D supplementation to improve the vitamin D status of breast-fed infants: a randomized controlled trial. Mayo Clin Proc. 2013 Dec;88(12):1378-87. doi: 10.1016/j.mayocp.2013.09.012. PMID 24290111